CLINICAL TRIAL: NCT03117517
Title: Effects of Metformin and Combination of Metformin and Pioglitazone on Plasma Interleukin-6 and Interleukin-8 Levels in Polycystic Ovarian Syndrome
Brief Title: Treatment With Metformin and Combination of Metformin and Pioglitazone in Polycystic Ovarian Syndrome
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Responsible Party: Principal Investigator, Mohsin Shah, Assistant Professor, Khyber Medical University Peshawar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Protocol KMU/CTU/2016/02
Record Dates: First submitted 2017-03-21; First posted 2017-04-18 (Actual); Results first posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Polycystic Ovarian Syndrome
Keywords: PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin; Pioglitazone

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Experimental): Drug intervention: Metformin 500 mg tablet twice orally for 3 months
  Interventions: Drug: Metformin
- Metformin, pioglitazone (Active Comparator): Drugs intervention: Combination of Metformin (1000 mg) and pioglitazone (30 mg) tablets will be given orally for 3 months
  Interventions: Drug: Metformin, Pioglitazone

INTERVENTIONS:
Drug: Metformin — Metformin (1000 mg)
  Other Names: Glucophage
  Arms: Metformin
Drug: Metformin, Pioglitazone — Metformin (1000 mg) Pioglitazone (30 mg)
  Other Names: Glucophage, Zolid
  Arms: Metformin, pioglitazone

SUMMARY:
Objective:

1. To investigate the changes in the levels of interleukin-6 and interleukin-8 after 3 months treatment with metformin alone and combination of metformin and pioglitazone in patients with polycystic ovarian syndrome (PCOS).
2. To evaluate insulin resistance in all the groups at baseline and after 3 months of treatment.

Design: Two-Arm Randomized Clinical trial.

Setting: Out-Patient Department (OPD) of Mardan Medical Complex, Khyber Medical University.

Patient(s): One hundred and two patients with PCOS.

Intervention(s): 51 women will receive metformin according to the body weight with maximum dose of 1000 mg (BD) daily. Remaining 51 will receive metformin and pioglitazone combination according to the body weight with maximum dose of 1000 mg and 30 mg (BD) daily.

Main outcomes measure(s): Serum concentrations of fasting blood glucose, insulin, homeostatic model assessment for insulin resistance (HOMA-IR), follicle stimulating hormone (FSH), luteinizing hormone (LH), interleukin-6 (IL-6) and i-nterleukin-8 (IL-8).

DETAILED DESCRIPTION:
Effects of metformin and combination of metformin and pioglitazone on plasma IL-6 and IL-8 levels in polycystic ovarian syndrome

Sponsor:

Office of Research, Innovation and Commercialization (ORIC)

Khyber Medical University (KMU), Peshawar, Pakistan

Hayatabad, Phase 5.

Collaborations:

This study is a collaborative project between Khyber Medical University Peshawar; Mardan Medical Complex, Mardan and Department of Human Pathology in Adulthood and Childhood "Gaetano Barresi", University of Messina (Italy).

Coordinating Center:

Clinical Trial Unit (CTU), Khyber Medical University, Peshawar

Pakistan

Email: CTU@kmu.edu.pk

Study Chair

Dr. Mohsin Shah

Collaborative Group Chairs

Dr. Farhat Rehman, Dr. Salvatore Giovanni Vitale M.D.

CTU KMU Staff:

Clinical Lead: Dr. Asif Ali

Statistician: Dr. Muhammad Naseem/Dr. Zia Ul Haq

Project Manager: Dr. Mohsin Shah, Dr. Dur-e- Shehwar Ali

Emergency contact:

Name: Dr. Farhat Rehman; Phone: 0301 8192880

1. Introduction:

   Polycystic ovarian syndrome (PCOS) is a common endocrinopathy affecting women of reproductive age, with a frequency of about 4 to 7% (11). The syndrome is characterized by chronic oligo-anovulation, polycystic ovaries and hyperandrogenism (1). The patient has signs and symptoms of infertility, increased risk of insulin resistance, irregular menstruation (oligo-amenorrhea), hyperinsulinemia, type II diabetes mellitus, insulin resistance, increase hair growth (1).

   Metformin, basically a biguanide, is an anti-hyperglycemic agent that improves glucose tolerance, increases the action of insulin at cellular levels without affecting insulin secretion (2). Metformin has been used in the management of insulin resistance, hyperinsulinemia and lipid abnormalities (2). A positive effect of metformin is proved by several studies on both metabolic and reproductive aspects in PCOS women (9). Metformin reduces obesity and decreases serum c-reactive protein levels in PCOS women (10). Pioglitazone is a thiazolidinedione (TZD) with hypoglycemic (anti-hyperglycemic, antidiabetic) action in the management of diabetes. It is also useful for reducing the cardiovascular risks associated with polycystic ovarian syndrome, having both anti-inflammatory and anti-arteriosclerotic properties (3). Pioglitazone was suggested to reduce the incidence of diabetes mellitus by more than 50% with administration of pioglitazone in PCOS (3). Interestingly, the protection from developing diabetes mellitus in these patients remained even when pioglitazone was stopped (3).

   IL-6, a major pro-inflammatory cytokine, shows an essential part in endocrine system, particularly related to ovarian growth and the course of fertilization and implantation (1). IL-6 plays an important role in facilitating low grade chronic inflammation in patients with PCOS (1). IL-6 has been shown to be closely related to insulin resistance and cardiovascular abnormalities (4). Obesity, a major risk factor for type II diabetes, was reported to be associated with elevated IL-6 levels (4).

   IL-8 is a chemokine formed via macrophages and other cell types like endothelial cells, airway smooth muscle cells and epithelial cells (6). The levels of IL-6 and IL-8 were decreased in patients of PCOS after they reduced their insulin resistance and body weight (4). The manifestation of increased markers such as c-reactive protein, IL-6, IL-8 levels and raised leukocyte count is indication of low grade inflammation in women with PCOS (8). Elevated levels of IL-6 and IL-8 were related with an increased risk of atherosclerosis and future myocardial infarction (4).

   The investigators designed this study to elucidate the role of metformin and combination of metformin and pioglitazone in reducing the levels of IL-6 and IL-8 in patients with PCOS. The study will help in deciding a better treatment regimen for patients with PCOS. IL-6 and IL-8 may emerge as predictive biomarkers of treatment response.
2. Aims and objectives

Objectives:

The objectives of this study are

1. Primary

   To investigate the changes in the levels of IL-6 and IL-8 after 3 months treatment with metformin alone and combination of metformin and pioglitazone in patients with PCOS.
2. Secondary

   To evaluate insulin resistance in all the groups at baseline and after 3 months of treatment.
3. Hypothesis:

Combination of metformin and pioglitazone may decrease the levels of IL-6 and IL-8 in women with PCOS better than metformin.

5. Materials and Methods:

1. Study design: Two-Arm Randomized Clinical trial.
2. Study settings: Out-Patient Department (OPD) of Mardan Medical Complex, Khyber Medical University
3. Study duration: Six Months after approval of proposal
4. Sample size:

   The sample size was calculated using OpenEpi software. With an expected reduction in IL-6 and IL-8 values of 15% in the metformin arm, the investigators would need 102 women with PCOS to demonstrate a 40% reduction in IL-6 and IL-8 in the metformin and pioglitazone arm with a power of at least 80% and a ratio of 1 in the two arms.

   Arm#1: 51 women with PCOS will be selected based on the inclusion and exclusion criteria. The participants will receive metformin according to the body weight with maximum dose of 1000 mg (BD) daily.

   Arm#2: 51 women with PCOS will be selected based on the inclusion and exclusion criteria. The participants will receive metformin and pioglitazone combination according to the body weight with maximum dose of 1000 mg and 30mg (BD) daily.
5. Sampling techniques: Blood samples will be taken from ante cubital vein after an overnight fast. Samples will be taken from all groups at the initiation and at the end of 3 months. Serum levels luteinizing hormone (LH), follicle stimulating hormone (FSH), prolactin, testosterone, IL-6, IL-8 and insulin will be analyzed by ELISA method. Fasting glucose will be performed by chemistry analyzer. Evaluation of insulin resistance will be performed by using HOMA-IR Index (Homeostasis model assessment for insulin resistance) with following formula. :

   HOMA-IR= fasting plasma insulin (µIU/mL) x fasting plasma glucose (mmol/L) /22.5

   6. Subject Population:

   6.1 Target population

   Women with PCOS visiting the outpatient department of participating hospitals.

   6.2 Sample selection:

   Participants will be recruited in the study based on inclusion and exclusion criteria.

   6.3 Screening:

   Before the study-specific screening and investigations, patient will sign a written informed consent and the investigator will also sign the consent with date.

   6.4 Registration:

   Subjects will be registered before starting study treatment and a registration number will be allotted. Requests for registration will only be accepted from authorized investigators at sites that have received ethical approval. Treatment would be planned to start after registration. Registration would be done according to the instructions in the protocol only after all screening assessments have been performed and the responsible investigator has both verified the subject's eligibility and signed the completed registration form.

   Once the registration process has completed as per the instructions in the protocol, the subject will be assigned a subject, study number, and written confirmation of registration will be provided to the site. Individuals must be registered once in this trial.

   6.5 Randomization:

   Randomization will be performed using Block Randomization technique using online software Sealed Envelope.

   7. Data Collection Procedure:

   7.1 Patient Recruitment:

   Approval of the study will be obtained from the Khyber Medical University, Ethics Board. Potential participants will be identified in the participatory center. Purpose and components of the study will be explained to each potential participant. Once the participant has agreed to take part, the participant will be screened for eligibility criteria. All eligible participants will be asked to give a written informed consent. Data regarding age, weight, height, menstrual irregularity, hirsutism, past medical and surgical history, serum testosterone and fasting insulin will be taken. Each participant will undergo ultrasound for assessment of ovarian changes. The study participants will be grouped in the following two arms.

   Arm#1: 51 women with PCOS will be selected based on the inclusion and exclusion criteria. The participants will receive metformin according to the body weight with maximum dose of 1000 mg (BD) daily.

   Arm#2: 51 women with PCOS will be selected based on the inclusion and exclusion criteria. The participants will metformin and pioglitazone according to the body weight with maximum dose of 1000 mg and 30 mg (BD) daily.

   Arm 1 metformin (1000 mg)

   Arm 2 metformin (1000 mg)

   and pioglitazone (30 mg)

   7.2 Concomitant medication reporting and treatment:

   Concomitant medications will not be recorded during the study. The following medications and treatment are recommended during the study.

   7.2.1 Permitted

   The following medications are permitted during the study: Nonsteroidal Antiinflammatory Drugs (NSAIDs), multivitamins, antibiotics and proton pump inhibitors (PPIs).

   7.2.2 Use with caution

   There are no medications that should specifically be used with caution in this study.

   7.2.3 Prohibited

   There are no medications and treatments that are specifically prohibited in this study.

   7.2.4 Compliance

   Subject medication compliance will be determined at each visit after 1 month and the patient will be counseled appropriately if significant non-compliance is determined.

   7.2.5 Treatment discontinuation

   The treatment of the patient or study on the subject will be discontinued in case of pregnancy or any disease given in exclusion criteria and in patient with hypersensitivity to drugs. There is no serious adverse effect observed after treatment discontinuation.

   Data Analysis Procedure:

   Mean ± SD will be used for numeric data generated from our work. In each arm the mean difference in the IL-6 and IL-8 values will be calculated using paired sample t test. For between arms analysis, mean difference in the IL-6 and IL-8 values will be calculated using independent sample t test. Non-parametric statistics will be used if the data is skewed. A cut-off will be calculated for IL-6 and IL-8 separately using ROC curve analysis. Based on the cut-off, a binary logistic regression analysis will be performed to evaluate the predictive significance of the two treatment arms in reducing the levels of inflammatory markers IL-6 and IL-8. P-value of < 0.05 will be considered significant. Results will be presented in form of tables & figures. Statistical Package for the Social Sciences (SPSS), version 21 will be used for all the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed patients of PCOS.
* Must Swallow the tablet(s).
* Must give informed consent.

Exclusion Criteria:

* Women with cushing syndrome, hyperprolactinemia.
* Late onset congenital adrenal hyperplasia, androgen-producing tumors, pregnancy.
* Insulin dependent diabetes.
* Thyroid disease.
* Medications that alters the biochemical or hormonal profile.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — PCOS women with oligo-anovulation, hirsutism, elevated serum testosterone levels, menstrual cycle irregulary.
Enrollment: 106 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-08-29 (Actual); Study Completion 2018-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohsin Shah, PhD, Principal Investigator — Institute oF Basic Medical Sciences
Locations (1):
- Mardan Medical Complex, Mardan, Khyber Pukhtunkhwah, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The data collected at baseline and after treatment with metformin alone for 3 months which is ARM #1 in this study and treatment of patients with combination of metformin and pioglitazone which is ARM # 2 in this study for three months. Blood samples will be collected and processed for analysis. All the data collected from these patients at baseline and after 3 months of treatment will be available to other researchers in the form of publication and rest of the materials can be obtained from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: March 31, 2018 for next 5 years
Access Criteria: Publication

REFERENCES:
- [Background] Peng Z, Sun Y, Lv X, Zhang H, Liu C, Dai S. Interleukin-6 Levels in Women with Polycystic Ovary Syndrome: A Systematic Review and Meta-Analysis. PLoS One. 2016 Feb 5;11(2):e0148531. doi: 10.1371/journal.pone.0148531. eCollection 2016. PMID 26849353
- [Background] Ortega-Gonzalez C, Luna S, Hernandez L, Crespo G, Aguayo P, Arteaga-Troncoso G, Parra A. Responses of serum androgen and insulin resistance to metformin and pioglitazone in obese, insulin-resistant women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2005 Mar;90(3):1360-5. doi: 10.1210/jc.2004-1965. Epub 2004 Dec 14. PMID 15598674
- [Result] Xu X, Du C, Zheng Q, Peng L, Sun Y. Effect of metformin on serum interleukin-6 levels in polycystic ovary syndrome: a systematic review. BMC Womens Health. 2014 Aug 5;14:93. doi: 10.1186/1472-6874-14-93. PMID 25096410
- [Result] Velazquez EM, Mendoza S, Hamer T, Sosa F, Glueck CJ. Metformin therapy in polycystic ovary syndrome reduces hyperinsulinemia, insulin resistance, hyperandrogenemia, and systolic blood pressure, while facilitating normal menses and pregnancy. Metabolism. 1994 May;43(5):647-54. doi: 10.1016/0026-0495(94)90209-7. PMID 8177055
- [Result] Palomba S, Falbo A, Chiossi G, Orio F, Tolino A, Colao A, La Sala GB, Zullo F. Low-grade chronic inflammation in pregnant women with polycystic ovary syndrome: a prospective controlled clinical study. J Clin Endocrinol Metab. 2014 Aug;99(8):2942-51. doi: 10.1210/jc.2014-1214. Epub 2014 May 29. PMID 24873996

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metformin | Metformin, Pioglitazone
Started | 53 | 53
Completed | 48 | 49
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Metformin, Pioglitazone | Total
Number analyzed (Participants) | 53 | 53 | 106
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.63 (4.55) | 25.44 (3.74) | 25.53 (6.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 53 | 106
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — Population: Participants drop-out in follow-up.
  Participants
    Pakistan | 53 | 53 | 106

OUTCOME MEASURES:

1. Primary Outcome: Cytokines and Chemokines Measurements
Description: IL-6 and IL-8 levels by ELISA method using commercially available kits.
Time Frame: Baseline and after 3 Months
Population: Measurement of IL-6 levels in serum samples at baseline and after 3 months of treatment
Measure: Geometric Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Metformin | Metformin, Pioglitazone
Number analyzed (Participants) | 53 | 53
pg/ml
  IL-6 levels at baseline | 14.60 [12.05 to 17.69] | 14.12 [11.58 to 17.23]
  IL-6 levels after 3 months of treatment | 12.65 [10.61 to 15.08] | 11.12 [10.02 to 12.33]
  IL-8 Llevels at baseline | 61.92 [52.95 to 72.41] | 41.86 [38.24 to 45.83]
  IL-8 Llevels after treatment | 32.70 [22.99 to 46.50] | 22.00 [16.76 to 28.88]

2. Secondary Outcome: Hormonal Profiles
Description: Serum level of LH was measure at baseline and after 3 months of treatment
Time Frame: Baseine and after 3 Months
Population: Serum LH level at basline
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/ml
Groups:
- Metformin: Drug intervention: Metformin 500 mg tablet twice orally for 3 months
  Metformin: Metformin (1000 mg)
  Serum level of LH, FSH and testosterone
- Metformin, Pioglitazone: Drugs intervention: Combination of Metformin (1000 mg) and pioglitazone (30 mg) tablets will be given orally for 3 months
  Metformin, Pioglitazone: Metformin (1000 mg) Pioglitazone (30 mg)
  Serum level of LH, FSH and testosterone
Arm/Group | Metformin | Metformin, Pioglitazone
Number analyzed (Participants) | 53 | 53
mIU/ml
  LH level at baseline | 5.79 [4.95 to 6.77] | 6.625 [5.52 to 7.94]
  LH level after treatment | 4.92 [4.33 to 5.59] | 5.16 [4.50 to 5.91]

3. Secondary Outcome: Insulin Resistance
Description: Insulin resistance was measure by calculating HOMA-IR from the data of insulin and sugar levels.
Time Frame: Baseline and after 3 months
Population: Insulin resistance was determined by HOMA-IR
Measure: Mean (Standard Deviation); unit: unitless
Groups:
- Metformin: Drug intervention: Metformin 500 mg tablet twice orally for 3 months
  Metformin: Metformin (1000 mg)
  HOMA-IR at baseline and after treatment
- Metformin, Pioglitazone: Drugs intervention: Combination of Metformin (1000 mg) and pioglitazone (30 mg) tablets will be given orally for 3 months
  Metformin, Pioglitazone: Metformin (1000 mg) Pioglitazone (30 mg) HOMA-IR at baseline and after treatment
Arm/Group | Metformin | Metformin, Pioglitazone
Number analyzed (Participants) | 53 | 53
unitless
  HOMA-IR at baseline | 7.19 (3.00) | 6.22 (2.65)
  HOMA-IR after treatment | 3.97 (2.03) | 3.84 (2.13)

ADVERSE EVENTS:
Description: The drug used in this trial is safe for use in human studies. All-Cause Mortality, Serious, and OtherAdverse Events were not monitored/assessed.
Arm/Group | Metformin | Metformin, Pioglitazone
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
No blinding No measure of visceral adiposity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT03117517/SAP_000.pdf
  • Study Protocol (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT03117517/Prot_001.pdf